CLINICAL TRIAL: NCT06942650
Title: The Effect of Prolonged ischemıa and Anesthetic Agents on oxıdatıve Stress Parameters, postoperatıve Pain, and Postoperative Analgesia Requirement
Brief Title: The Effect of Prolonged ischemıa and anesthetıc Agents on Oxidative Stress
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/02; Duzce University (Other: Duzce University scientific research projects department)
Record Dates: First submitted 2025-03-18; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Tourniquet Pain; Ischemia-reperfusion; Postoperative Pain; Anesthesia; Oxydative Stress
Keywords: Hypoxia-inducible factor alfa; tourniquet pain; anesthesia; ischemia; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the relationship between postoperative pain and tourniquet-induced oxidative damage in adults undergoing orthopedic knee arthroscopy surgery.The goal of this observational study is to learn about the relationship between postoperative pain and tourniquet-induced oxidative damage in adults undergoing orthopedic knee arthroscopy surgery.

The main question it aims to answer is:

Does anesthetic agents used will affect tourniquet-related oxidative stress and postoperative pain ?

DETAILED DESCRIPTION:
Approval was received from Duzce University Clinical Research Ethics Committee(Decision no: 2019/02). Düzce University Among the patients who applied to the Orthopaedics Clinic of Düzce University Medical Faculty, Research and Application Hospital's Orthopaedics Clinic, and planned a knee arthroscopy operation, 60 patients with ASA I-II status who accepted participation and signed the informed consent were included in the study after receiving general anaesthesia. 1 patient was excluded from the study in the analysis part. The results of a total of 59 patients were analysed.

Patients underwent routine anaesthetic examination during preoperative preparation. Informed consent was obtained from all patients. All patients were pressurised at a 90-degree angle to the knee with an algometer (J Tech Commender Echo Algometer, USA), and the average of three measurements was taken. The pressure was displayed in grams (gr) on the digital screen on the front of the devices. The first pressure value at which the patient felt pain was recorded in gr. Measurements were made at three levels (lower, middle, upper) 3-4 cm from the incision site. Measurements around the incision site

Patients were prepared for the operation according to the timing and conditions planned by the relevant clinic, and no preoperative or operative interventions were made regarding the method of operation or anesthesia. The oxidative load (HIF and DAF-16) [ Human hypoxia-inducible factor 1α(HIF-1α) ELISA kit (pg/L), Human decay-accelerating factor(DAF/CD55)ELISA (pg/L) ] was measured from the centrifuged blood. In routine practice for knee arthroscopy operation under general anesthesia; ECG, pulsoximetry (O2 level measurement with finger probe), blood pressure measurement with cuff, tissue oximetry (NIRS, tissue oxygenation evaluation with probe attached to the relevant skin surface - dorsum of the foot) , patient monitoring was provided and the operation was started by positioning the patients after general anesthesia induction. Blood samples were taken from the foot to be operated on before the tourniquet was inflated and opened. Oxidative stress parameters were analyzed. Within the scope of the study, blood pressure values were recorded in the preoperative period (T0), while the patients were lying flat on the back after general anesthesia (T1), 5 minutes after the tourniquet was placed on the leg to be operated and inflated (T2), 15 minutes later (T3), 30 minutes later (T4), 60 minutes later (T5), before the tourniquet was opened (T6), and after the tourniquet was opened (T7). Tourniquet application was performed as routine, 20 mmHg above the initial blood pressure value, and the tourniquet was lowered in 1 second at the end of the operation. After the tourniquet was removed, d slope time (desaturation descent time), RR time (resaturation ascent time), delta StO2 (difference in tissue oximetry values between before and after anesthesia), hyperemic peak value, hyperemic period time after ischemia were recorded on the tissue oximetry trend monitor (Figure 2). Tourniquet time, duration of operation, duration of anaesthesia, patient's age, weight, height, body mass index, total anaesthetic agent usage, total tramadol administered (24-hour patient-controlled analgesia), and anaesthetic agent doses were recorded. Blood pressure and tissue oximetry values were obtained. Routine awakening and analgesia protocols were applied to the patients. Postoperative pain scale (VAS), operated and non-operated knee algometer values were measured at 1 hour, 3 hours, 6 hours, 12 hours, and 24 hours after awakening. Demographic outcomes, anaesthetic agent amounts, pain scores, HIF-1 alpha, and DAF measurements were analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years,
* (American society of Anesthesiologist) ASA I-II status,
* undergoing knee arthroscopy.

Exclusion Criteria:

* Diabetes mellitus,
* advanced chronic obstructive pulmonary disease,
* liver failure,
* renal failure,
* history of previous bypass,
* hemoglobinopathies,
* anemia,
* hypertensive patients,
* neurodegenerative diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sixty patients aged 18-80, with ASA I-II status, who underwent knee arthroscopy were included in the study. A voluntary consent form was obtained all th e patients.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
To observe the relation between somatic oximeter values and oxidative stress parameters. | 1 day
  To observe the correlation between INVOS™ 5100C Cerebral/Somatic Oximeter measurements(rSO2) (% value) and oxidative stress parameters [ Human hypoxia-inducible factor 1α(HIF-1α) ELISA kit (pg/L), Human decay-accelerating factor(DAF/CD55)ELISA (pg/L) ] measurements after tourniquet inflation and before tourniquet deflation.

SECONDARY OUTCOMES:
The effect of anesthetic agents on oxidative stress parameters. | 1 day
  To investigate the correlation between deslurane (ml), sevoflurane (ml), penthotal(mg), and propofol(mg) usage (ml) to tourniquet-related oxidative stress parameters [Human hypoxia-inducible factor 1α(HIF-1α) ELISA kit (pg/L), Human decay-accelerating factor(DAF/CD55)ELISA (pg/L) ]

OTHER OUTCOMES:
The effect of oxidative stress parameters on 24 hour analgesic needing | 1 day
  To investigate the correlation between 24-hour tramadol (mg), paracetamol (mg), fentanyl (mcg), and remifentanyl (mcg) usage with oxidative stress parameters [ Human hypoxia-inducible factor 1α(HIF-1α) ELISA kit (pg/L), Human decay-accelerating factor(DAF/CD55)ELISA (pg/L) ]

CONTACTS AND LOCATIONS:
Overall Officials: İlknur S YORULMAZ, Assoc. Prof., Principal Investigator — Duzce University
Locations (1):
- İlknur SuidiyeYORULMAZ, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided